CLINICAL TRIAL: NCT05029908
Title: Evaluation of the Relationship Between Parafunctional Habits, Pain and Functional Limitation of the Jaw in Temporomandibular Disorders
Brief Title: the Relationship Between Parafunctional Habits, Pain and Functional Limitation of the Jaw
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Cansin Medin, principal investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: 2021/209
Record Dates: First submitted 2021-08-30; First posted 2021-09-01 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Temporomandibular Disorder; Pain, Joint
Keywords: temporomandibular disorder; oral behavioral checklist; DC/TMD
MeSH Terms: conditions — Temporomandibular Joint Disorders; Arthralgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TMD disorders: 75 patients with temporomandibular disorder (TMD) who will apply to the outpatient clinic of Istanbul Physical Therapy and Rehabilitation Training and Research Hospital will be included in our study. Ethics Committee approval was obtained from Bakırköy Sadi Konuk Training and Research Hospital before starting the study and a voluntary consent form will be signed by the patients before the evaluation.
  In this cross-sectional study; 75 participants aged 18-65 years who has temporomandibular joint (TMJ) complaints for more than 3 months and has the cognitive ability to understand test instructions will be included. Patients with a history of previous TMJ operation, muscle, neurological or rheumatic disease that may affect TMJ, and a history of facial/cervical trauma or neoplasia will excluded from the study.
  Interventions: Diagnostic Test: Jaw Functional Limitation Scale

INTERVENTIONS:
Diagnostic Test: Jaw Functional Limitation Scale — DC/TMD Axis I TMD Pain Screener Questionnaire and TMD Symptom Questionnaire will be administered to the participants. To determine parafunctional habits and limitation of function, the DC/TMD Axis II assessment tools 'Jaw Functional Limitation Scale-8 (JFLS-8) and Oral Behavioral Checklist (OBC) will be applied. In addition, demographic data (age, gender, education level, occupation) will be questioned.

SUMMARY:
Temporomandibular disorders affect the general health and quality of life of individuals by causing deterioration in orofacial function and cause functional limitation. The use of Diagnostic Criteria for Temporomandibular Disorders (DC-TMD) is recommended for evidence-based evaluation of jaw joint disorders for clinical and research purposes.The aim of this study is to show the factors affecting the functional limitation of the jaw and to evaluate the relationship between the pain, Oral Behavioral Checklist and the Jaw Functional Limitation Scale (JFLS-8), using the Diagnostic Criteria for Temporomandibular Disorders (DC-TMD).

75 patients with temporomandibular disorder (TMD) who will apply to the outpatient clinic of Istanbul Physical Therapy and Rehabilitation Training and Research Hospital will be included in our study.

DC/TMD Axis I TMD Pain Screener Questionnaire, TMD Symptom Questionnaire, DC/TMD Axis II assessment tools 'Jaw Functional Limitation Scale-8 (JFLS-8) and Oral Behavioral Checklist (OBC) will be applied. In addition, demographic data will be questioned.

DETAILED DESCRIPTION:
Temporomandibular disorders affect the general health and quality of life of individuals by causing deterioration in orofacial function and cause functional limitation. The use of Diagnostic Criteria for Temporomandibular Disorders (DC-TMD) is recommended for evidence-based evaluation of jaw joint disorders for clinical and research purposes.The aim of this study is to show the factors affecting the functional limitation of the jaw and to evaluate the relationship between the pain, Oral Behavioral Checklist and the Jaw Functional Limitation Scale (JFLS-8), using the Diagnostic Criteria for Temporomandibular Disorders (DC-TMD).

75 patients with temporomandibular disorder (TMD) who will apply to the outpatient clinic of Istanbul Physical Therapy and Rehabilitation Training and Research Hospital will be included in our study. Ethics Committee approval was obtained from Bakırköy Sadi Konuk Training and Research Hospital before starting the study and a voluntary consent form will be signed by the patients before the evaluation.

In this cross-sectional study; 75 participants aged 18-65 years who has temporomandibular joint (TMJ) complaints for more than 3 months and has the cognitive ability to understand test instructions will be included. Patients with a history of previous TMJ operation, muscle, neurological or rheumatic disease that may affect TMJ, and a history of facial/cervical trauma or neoplasia will excluded from the study.

DC/TMD Axis I TMD Pain Screener Questionnaire and TMD Symptom Questionnaire will be administered to the participants. To determine parafunctional habits and limitation of function, the DC/TMD Axis II assessment tools 'Jaw Functional Limitation Scale-8 (JFLS-8) and Oral Behavioral Checklist (OBC) will be applied. In addition, demographic data (age, gender, education level, occupation) will be questioned.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years
* temporomandibular joint complaints for more than 3 months
* cognitive ability to understand test instructions

Exclusion Criteria:

* history of previous temporomandibular joint operation, muscle, neurological or rheumatic disease that may affect temporomandibular joint
* history of facial/cervical trauma or neoplasia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 75 patients with temporomandibular disorder (TMD) who applied to the outpatient clinic of Istanbul Physical Therapy and Rehabilitation Training and Research Hospital will be included in our study.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2021-04-25 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Jaw Functional Limitation Scale | baseline
  Jaw Functional Limitation Scale-8 (JFLS-8)is a scale in the DC / TMD Axis II section and aims to evaluate the functional limitation of the jaw. It consists of eight items that assess restraint due to temporomandibular problems, and these include changes in jaw motility (item 4), chewing (items 1-3), and verbal and emotional expression. (item 5-8).

CONTACTS AND LOCATIONS:
Overall Officials: cansın m ceylan, Principal Investigator — istanbul physical medicine and rehabilitation research and training hospital
Locations (1):
- Cansın Medin Ceylan, Istanbul, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No